CLINICAL TRIAL: NCT05888753
Title: A Novel Study, Textbook Outcome in Adrenal Neoplasms: Observational Study in a Endocrine Surgical Unit.
Brief Title: Textbook Outcome in Adrenal Neoplasms
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Candido Fernando Alcazar-Lopez, Principal Investigator, Physician, Hospital General Universitario de Alicante
Other Study IDs: 05/2023
Record Dates: First submitted 2023-05-24; First posted 2023-06-05 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Outcome Assessment; Adrenal Neoplasm
MeSH Terms: conditions — Adrenal Gland Neoplasms | interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Yes Textbook Outcome: Patients undergoing scheduled adrenal neoplasm surgery with a R0 resection, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days
  Interventions: Procedure: Adrenalectomy
- No Textbook outcome: Patients undergoing scheduled colon cancer surgery without any of the following items: R0 resection, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days
  Interventions: Procedure: Adrenalectomy

INTERVENTIONS:
Procedure: Adrenalectomy — Scheduled adrenal surgery

SUMMARY:
BACKGROUND:

Textbook outcome (TO) is a multidimensional quality management tool that uses a set of traditional surgical measures to reflect an "ideal" surgical result for a particular pathology. The aim of the present study is to record the rate of TO in patients undergoing elective surgery for adrenal neoplasms.

MATERIAL AND METHODS:

Retrospective study of all patients undergoing scheduled adrenal neoplasms surgery at a Spanish university hospital from September January 2010 to December 2022. Emergency surgeries were excluded. The variables included in the definition of TO were: R0 resection, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days.

The main objective of this study is to analyse the achievement of TO in a series of patients undergoing scheduled adrenal neoplasms resection at the Doctor Balmis General University Hospital in Alicante, Spain. The investigators compare the group of patients who achieve a TO result with the group of patients who do not. A univariable and multivariable analysis will be carry out in order to indentified the variables associated with TO.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective adrenal resection were eligible for the study

Exclusion Criteria:

* Age under 18 years
* Emergency surgery
* Resections of other organs in the same surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective adrenal resection in the endorine surgical unit in public universitary hospital of alicante
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Textbook Outcome | January 2010 to December 2022
  Analyse the achievement of Textbook Outcome in a series of patients undergoing scheduled adrenal resection. Number of Participants with R0 resection, no Clavien-Dindo ≥IIIa complications, no prolonged stay (<P75), no readmissions, and no mortality in the first 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Jesús Rubio García, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rubio-Garcia JJ, Gil Navarro R, Franco Campello M, Costa Navarro R, Gomis Martin A, Villodre Tudela C, Zaragoza Zaragoza C, Carrion Tomas A, Ramia-Angel JM. A novel study, textbook outcome in adrenalectomy: retrospective observational study in an endocrine surgical unit. Updates Surg. 2024 Apr;76(2):565-571. doi: 10.1007/s13304-024-01756-z. Epub 2024 Feb 5. PMID 38316738